CLINICAL TRIAL: NCT01929941
Title: A Phase 1, Open-Label, Dose-Escalation, Safety and Tolerability Study of INCB047986 in Subjects With Advanced Malignancies
Brief Title: An Open-Label Study of a Novel JAK-inhibitor, INCB047986, Given in Patients With Advanced Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 47986-103
Record Dates: First submitted 2013-08-22; First posted 2013-08-28 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Solid Tumor; Hodgkin's Lymphoma; NHL (Non-Hodgkin Lymphoma); Pancreatic Cancer; Breast Cancer; UC (Ureter and Urethera); Advanced Cancer; Metastatic Cancer
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Pancreatic Neoplasms; Breast Neoplasms; Neoplasm Metastasis | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 INCB047986 (Experimental)
  Interventions: Drug: INCB047986
- Group 2 Experimental: INCB047986, gemcitabine, nab-paclitaxel (Experimental)
  Interventions: Drug: INCB047986; Drug: Gemcitabine; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: INCB047986 — Initial cohort dose of INCB047986 monotherapy at the protocol-specified starting dose, with subsequent cohort escalations based on protocol-specific criteria
  Arms: Group 1 INCB047986
Drug: INCB047986 — INCB047986 tablets administered orally at the protocol specified dose and frequency
  Arms: Group 2 Experimental: INCB047986, gemcitabine, nab-paclitaxel
Drug: Gemcitabine — Gemcitabine administered intravenously over 30 minutes at the protocol-specified dose and frequency
  Other Names: Gemzar®
  Arms: Group 2 Experimental: INCB047986, gemcitabine, nab-paclitaxel
Drug: nab-paclitaxel — nab-paclitaxel administered intravenously over 30 minutes at the protocol-specified dose and frequency
  Other Names: Abraxane®
  Arms: Group 2 Experimental: INCB047986, gemcitabine, nab-paclitaxel

SUMMARY:
This is an open-label study of INCB047986 given to two distinct groups of patients (Group 1 and Group 2) with advanced malignancies. The purpose of the study is to evaluate the safety, tolerability and pharmacokinetics of INCB047986 and to determine the maximum tolerated dose of INCB047986 in combination with gemcitabine and nab paclitaxel in a select group of patients with solid tumors. Each patient group will participate in a phase of the study which is divided into two parts. The patient groups will be enrolled in a sequential manner starting with Patient Group 1.

Patient Group 1

Group 1 will be comprised of patients with advanced malignancies who will receive INCB047986 as monotherapy.

Part 1: Dose Escalation Phase - This phase will evaluate the safety, tolerability and pharmacokinetics (PK) of INCB047986 when given as described to patients with advanced malignancies. A goal of Part 1 will be to identify the maximally tolerated dose (MTD) of INCB047986 and/or other dose(s) that are tolerated doses and produce a substantial pharmacologic effect. These doses will be used in Part 2 of the study.

Part 2: Expansion Phase - This phase will further explore the safety, tolerability, PK, and preliminary clinical activity of INCB047986 using the doses identified in Part 1.

Group 2

Group 2 will be in subjects with advanced or metastatic pancreatic cancer, breast cancer or urothelial cancer.

Part 1: Dose Optimization Phase - This phase will identify the MTD of INCB047986 in combination with gemcitabine and nab-paclitaxel in patients with advanced or metastatic solid tumors. Specifically, these will be patients with pancreatic adenocarcinoma (first or second line), triple-negative breast cancer (second line) or urothelial cancer (second line).

Part 2: Expansion Phase - This phase will explore the safety, tolerability, PK, biomarkers, and preliminary clinical activity of the dose regimen(s) identified in Part 1. Patients enrolled in this phase will be limited to those with advanced or metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

Group 1

* Aged 18 years or older, with histologically or cytologically confirmed solid tumor, Hodgkin's lymphoma, aggressive or indolent non-Hodgkin's lymphoma. (NOTE: Patients with acute and chronic leukemia, Burkitt's lymphoma, precursor B lymphoblastic leukemia/lymphoma, and myeloma are excluded)
* Life expectancy of 12 weeks or longer.
* Subject must have received ≥ 1 prior treatment regimen.
* The subject must not be a candidate for potentially curative therapy, including transplant.

Group 2

* Aged 18 years or older
* Part 1 - Histologically or cytologically confirmed pancreatic adenocarcinoma (first or second line), triple-negative breast cancer (second line), or urothelial cancer (second line)
* Part 2 - Histologically or cytologically confirmed pancreatic adenocarcinoma
* No more than 1 prior chemotherapy regimen for advanced or metastatic disease (not including neoadjuvant and/or adjuvant therapy).
* There is no restriction on the number of prior non-myelosuppressive targeted therapies or hormonal agents (e.g., epidermal growth factor receptor-targeted therapy for lung cancer and hormonal therapy for breast cancer or ovarian cancer); NOTE: Targeted and/or hormonal therapy alone will not be considered chemotherapy for the purposes of this study.

Exclusion Criteria:

Group 1 and 2

* Received an investigational study drug within 28 days or 5 half-lives (whichever is longer) prior to receiving their first dose of study drug.
* Received any approved anticancer medications within 21 days or 5 half-lives (whichever is longer) prior to receiving the first dose of study drug (42 days for nitrosoureas) EXCEPT steroids at ≤ 10 mg prednisone daily (or equivalent).
* Has any unresolved toxicity ≥ Grade 2 from previous anticancer therapy without medical monitor approval.

  o Subjects with ongoing chronic toxicities such as fatigue or neuropathy may be allowed after approval from the sponsor's medical monitor
* Evidence of uncontrolled brain metastases or history of spinal cord compression, or primary central nervous system (CNS) tumors.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of ≥ 2.
* Received allogeneic hematopoietic stem cell transplant within the last 6 months, or has active graft versus host disease (GVHD) following allogeneic transplant, or is currently receiving immunosuppressive therapy following allogeneic transplant.
* Received autologous hematopoietic stem cell transplant within the last 3 months.
* Radiation treatment within the previous 4 weeks.
* History of active hepatitis or positive serology for hepatitis B (unless due to vaccination) or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Adverse events that are defined as dose limiting toxicities occurring in the first 21 days of treatment in Group 1 and the first 28 days of treatment in Group 2. | Approximately 21 days (Group 1); Approximately 28 days (Group 2)
Safety and tolerability of INCB047986 monotherapy and in combination with gemcitabine and nab-paclitaxel as assessed by summary of clinical laboratory assessments, Electrocardiogram (ECG), and Adverse Events (AEs). | Group 1 and Group 2: up to 6 months
  Group 1: Baseline and weekly for Cycle 1 and then Day 1 for all subsequent cycles until the End of Treatment visit. Group 2: Baseline and weekly for Cycle 1 and then Day 1, Week 8 and Week 15 for all subsequent cycles until the End of Treatment visit.

SECONDARY OUTCOMES:
Tumor response rates will be derived from investigator assessment of response in subjects with measurable disease | Approximately 6 months
Plasma concentrations will be used to estimate peak plasma concentration (cmax) and area under the plasma concentration curve (AUC) | Day 15 of treatment at a given dose
Duration of Response (DOR) and Progression Free Survival (PFS) in subjects with measureable disease | Approximately 6 months
Plasma concentration of biomarkers and cytokines before and during treatment | Approximately 6 months
Change in body weight | Approximately 6 months
Change in Eastern Cooperative Oncology Group (ECOG) status from baseline to each visit where the variable is measured | Approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: William Williams, M.D., Study Director — Incyte Corporation
Locations (3):
- United States (3):
  - Atlanta, Georgia
  - Nashville, Tennessee
  - Dallas, Texas